CLINICAL TRIAL: NCT02475759
Title: Nutritional Prehabilitation Program and Cardiac Surgery Outcome in Pediatrics. A Randomized Controlled Trial
Brief Title: Nutritional Prehabilitation Program and Cardiac Surgery Outcome in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Ali El-Farrash, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASU 015
Record Dates: First submitted 2015-03-10; First posted 2015-06-19 (Estimated); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- two weeks prehabilitation group (Active Comparator): Nutritional perioperative prehabilitation program for two weeks in malnourished congenital heart disease children
  Interventions: Dietary Supplement: Nutritional perioperative prehabilitation program for two weeks
- one week prehabilitation group (Active Comparator): Nutritional perioperative prehabilitation program for one week in malnourished congenital heart disease children
  Interventions: Dietary Supplement: Nutritional perioperative prehabilitation program for one week

INTERVENTIONS:
Dietary Supplement: Nutritional perioperative prehabilitation program for two weeks — nutritional intervention received two weeks before surgical intervention
  Other Names: Nutritional perioperative prehabilitation program
  Arms: two weeks prehabilitation group
Dietary Supplement: Nutritional perioperative prehabilitation program for one week — nutritional intervention received one weeks before surgical intervention
  Other Names: Nutritional perioperative prehabilitation program
  Arms: one week prehabilitation group

SUMMARY:
Nutritional Prehabilitation Program and Cardiac Surgery Outcome in Pediatrics. A randomized controlled trial.

DETAILED DESCRIPTION:
Nutritional Prehabilitation Program and Cardiac Surgery in Pediatrics. A randomized controlled trial to compare the outcome of malnourished congenital heart surgery patients who randomly received nutritional rehabilitation program 2 weeks and 1 week before surgical intervention.

ELIGIBILITY:
The study included all infants with CHD, admitted to the cardiothoracic unit for either palliative or corrective surgery, and suffering from nutritional deficiencies with moderate or severe malnutrition .

Infants received long-term nutritional prehabiliatation. Those with congenital or acquired anomaly of the gastrointestinal tract; multiple congenital anomalies; chromosomal, metabolic,or endocrine diseases; any systemic illness; or fever or infection within 1 wk before the study entry were excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
daily feeding characteristics | admission
  daily feeding characteristics
anthropometric and laboratory measure | admission
  anthropometric and laboratory measure

SECONDARY OUTCOMES:
length of ICU stay | 3weeks
  length of ICU stay
duration of mechanical ventilation and extubation timing | 3 weeks
  total days of mechanical ventilation
postoperative vital stability, surgical complication,nosocomial sepsis,inotropes withdrawal | admission
  same as above

CONTACTS AND LOCATIONS:
Locations (1):
- 38 abbasia, next to nour mosque, Ain Shams University Hospital, Pediatrics department, Cairo, Egypt